CLINICAL TRIAL: NCT05879484
Title: A Phase Ib/II Multicenter Study of Front Line Pembrolizumab and Valemetostat in PD-L1 Positive, HPV-Negative Recurrent/Metastatic Squamous Cell Carcinoma (SCC) of the Head and Neck: The PANTHERAS
Brief Title: Study of Front Line Pembrolizumab and Valemetostat in PD-L1 Positive, HPV-Negative Recurrent/Metastatic Squamous Cell Carcinoma (SCC) of the Head and Neck: The PANTHERAS
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was never opened for enrollment as the CRADA was never executed
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 10001545; 001545-C
Record Dates: First submitted 2023-05-26; First posted 2023-05-30 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Sinonasal Cancer; Squamous Non-small Cell Lung Cancer; Lung Cancer; Head and Neck Squamous Cell Carcinoma; Head and Neck Carcnimona; Head and Neck Cancer
Keywords: Pd-L1 Inhibitor; Valemetostat + pembrolizumab; Pembrolizumab; Valemetostat
MeSH Terms: conditions — Lung Neoplasms; Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Pembrolizumab + de-escalating doses of valemetostat
  Interventions: Drug: pembrolizumab; Drug: valemetostat
- Arm 2 (Experimental): RP2D of valemetostat in combination with pembrolizumab
  Interventions: Drug: pembrolizumab; Drug: valemetostat

INTERVENTIONS:
Drug: pembrolizumab — Phase Ib: Pembrolizumab 200mg will be administered by IV infusion every 3 weeks.
  Phase II: Pembrolizumab 200mg will be administered by IV infusion every 3 weeks.
Drug: valemetostat — Phase Ib: Valemetostat will be given orally every day of every cycle (DL-1: 100mg, DL1: 150mg, DL2: 200mg).
  Phase II: Valemetostat will be given orally daily at the recommended phase 2 dose.

SUMMARY:
Background:

Head and neck squamous cell carcinoma (HNSCC) is the 6th most common cancer worldwide. These cancers have different causes, with smoking/tobacco exposure and human papilloma virus infection being the most common. . When HNSCC occurs in people who are not infected with HPV, the cancers are more likely to return after treatment; when this happens, overall survival is only about 10 months, thus better treatments are needed.

Objective:

To test a combination treatment using 2 drugs (valemetostat and pembrolizumab) in people with HNSCC. Phase 1b of the study will determine a recommended dose of the 2 drugs and evaluate how safe the combination is.; this will include patients with HPV-positive and HPV-negative HNSCC, as well as squamous cell NSCLC that have progressed on anti-PD-1/anti-PD-L1 therapies.Phase II will determine how effective the combination is and will focus on patients with HPV-negative HNSCC.

Eligibility:

People aged 18 years and older with HPV-negative HNSCC, sinonasal carcinoma of the head and neck, or squamous non-small cell lung cancer (NSCLC).

Design:

Participants will be screened. They will have a physical exam. They will have blood and urine tests and tests of their heart function. They will have imaging scans. They may have a biopsy: A small sample of tissue will be removed from the tumor.

Treatment will be given in 21-day cycles.

Pembrolizumab is administered through a tube attached to a needle inserted into a vein in the arm. Participants will receive pembrolizumab on the first day of each cycle.

Valemetostat is a tablet taken by mouth. Participants will take the tablet once a day at home. They will record the date and time of each dose in a diary. They will also write down any adverse effects they experience.

Participants may remain in the study up to 2 years.

DETAILED DESCRIPTION:
Background:

* Head and neck squamous cell carcinoma (HNSCC) is the 6th most common cancer worldwide, with approximately 60,000 patients diagnosed annually in the United States.
* Only 14% of HNSCC patients have structural defects in the genes encoding for the human leukocyte antigens (HLA) class I components, while a higher percentage of these tumors show downregulation of HLA class I components by immunohistochemistry supports those epigenetic mechanisms may be involved in the deregulation of these genes.
* Valemetostat (DS-3201) is an enhancer of zeste homolog 1 and 2 (EZH1/2) dual inhibitor that is actively being investigated in phase I and II trials for hematologic malignancies and is approved for adult T-cell leukemia/lymphoma (ATL) indication in Japan.
* Patients with recurrent or metastatic (R/M) pembrolizumab-na(SqrRoot) ve human papillomavirus (HPV)-negative HNSCC have a low 6-month progression-free survival (PFS) (28%) with pembrolizumab monotherapy, thus novel interventions are needed to increase the efficacy of pembrolizumab.

Objectives:

Phase Ib:

* To determine the recommended phase II dose (RP2D) of valemetostat in combination with pembrolizumab.
* To evaluate the safety of valemetostat in combination with pembrolizumab.

Phase II:

-To determine the disease control rate (DCR)=partial response (PR) + complete response (CR) + stable disease (SD).

Eligibility:

-Participants must have a diagnosis of locoregionally recurrent or metastatic (R/M) HPVnegative (Phase Ib and Phase II) or positive HNSCC (Phase Ib only): oral cavity, tonsil, pharynx, hypopharynx, larynx. Note: Nasopharyngeal carcinoma and cutaneous squamous cell carcinoma (SCC) are excluded

OR

(R/M) squamous non-small cell lung cancer (NSCLC) (Phase Ib only)

OR

(R/M) sinonasal carcinomas of the head and neck (Phase Ib only).

* Age >18 years.
* Adequate organ and marrow function.

Design:

* This is an open-label multicenter phase Ib/II study to evaluate the safety and efficacy of the combined treatment of valemetostat and pembrolizumab.
* During phase Ib we will estimate the RP2D of the valemetostat in combination with pembrolizumab.
* During phase II we will examine the efficacy and continue to evaluate the safety of the study regimen at the RP2D of the valemetostat in combination with pembrolizumab.
* Participants will receive treatment in cycles consisting of 21 (+/- 3) days for 2 years.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Participants must have a diagnosis of one of the following types of cancer:

   Phase Ib (Part A):

   -Histologically or cytologically confirmed locoregionally recurrent or metastatic (R/M) human papillomavirus (HPV)-negative* or -positive* squamous cell carcinoma of the head and neck: oral cavity, tonsil, pharynx, hypopharynx, larynx. Note: Nasopharyngeal carcinoma and cutaneous squamous cell carcinoma (SCC) are excluded.

   OR

   -Histologically or cytologically confirmed R/M sinonasal carcinomas of the head and neck.

   OR

   -Histologically confirmed R/M squamous non-small cell lung cancer (NSCLC).

   *HPV status will be determined by history of p16 IHC staining conducted per standard of care.

   Phase II (Part B):

   -Histologically or cytologically confirmed locoregionally R/M HPV-negative* squamous cell carcinoma of the head and neck: oral cavity, tonsil, pharynx, hypopharynx, larynx. Note: Nasopharyngeal carcinoma and cutaneous SCC are excluded.

   *HPV status will be determined by history of p16 IHC staining conducted per standard of care.
2. PD-L1 combined positive score (CPS) >= 1, confirmed by Food and Drug Administration (FDA) approved 22C3 PharmDx test.
3. Phase Ib only: Participants may be na(SqrRoot) ve or refractory to pembrolizumab or other PD- L1/PD-1 checkpoint inhibitors and may have had any number of lines of systemic therapy.
4. Phase II only: Participants must be pembrolizumab-naive and not have received PD- L1/PD-1 checkpoint inhibitors and must not have had prior lines of systemic chemotherapy or immunotherapy for recurrent or metastatic HNSCC.
5. Age >=18 years.
6. Eastern Cooperative Oncology Group (ECOG) performance status <=2 (Phase Ib) or <= 1 (Phase II).
7. Participants must have adequate organ and marrow function as defined below:

   7.1 Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <=3.0 X upper limit of normal (ULN)

   7.2 Total bilirubin <=1.5 X ULN. Note: Participants with Gilbert's syndrome may have total bilirubin <3.0 mg/dL

   7.3 Absolute neutrophil count (ANC) >=1.5 X 10^9/L

   7.4 Hemoglobin (Hgb) >=8.5 g/dL

   7.5 Platelet count >=75 X 10^9/L

   7.6 Creatinine clearance >=60 mL/min (calculated by the Cockcroft-Gault equation).
8. Acute non-hematologic toxic effects (as evaluated by NCI Common Terminology Criteria for Adverse Events (CTCAE), version 5.0 of any prior therapy (except alopecia) resolved as shown below:

   8.1 Peripheral motor neuropathy, Peripheral sensory neuropathy: Grade <=2

   8.2 Fatigue: Grade <=2

   8.3 All others: Grade <=1
9. Participants with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression within 4 weeks before study treatment initiation.
10. Participants with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate CNS specific treatment is not required per Standard of Care.
11. Participants must have measurable disease by RECIST 1.1.
12. Human immunodeficiency virus (HIV)-infected participants on effective anti-retroviral therapy with undetectable viral load are eligible for this trial.
13. For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated. Participants with a history of current HCV infection who are currently on treatment must have an undetectable HCV viral load to be eligible.
14. Women of child-bearing potential (WOCBP) must agree to use a highly effective method of contraception (hormonal, intrauterine device (IUD), surgical sterilization, abstinence) for the duration of the study treatment and up to 4 months after the last dose of the study drug(s).

    A female is considered of childbearing potential following menarche and until becoming postmenopausal (no menstrual period for a minimum of 12 months) unless permanently sterile (undergone a hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) with surgery at least 1 month before the first dose of study drug(s) or confirmed by follicle-stimulating hormone (FSH) test >40 mIU/mL and estradiol <40 pg/mL (<140 pmol/L).

    Men must agree to use an effective method of contraception (barrier, surgical sterilization, abstinence) for the duration of the study treatment and up to 4 months after the last dose of the study drug(s). We also will recommend men with female partners of childbearing potential to ask female partners to be on highly effective birth control (hormonal, intrauterine device (IUD), surgical sterilization).
15. Female participants must not donate, or retrieve for their own use, ova from the time of study treatment initiation and throughout the study treatment period, and for at least 4 months after the final study drug(s) administration. Male participants must not freeze or donate sperm within the same period.
16. Breastfeeding participants must be willing to discontinue breastfeeding from study treatment initiation through 4 months after the last dose of the study drug(s).
17. Participants must have disease amenable for biopsies (not used for evaluation of disease per RECIST 1.1) and be willing to undergo these biopsies (Phase II only).
18. The ability of a participant to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

1. History of allergic reactions attributed to compounds of similar chemical or biologic composition to valemetostat or pembrolizumab used in the study.
2. Prior curative radiation therapy or major surgery within 4 weeks or palliative radiation therapy within 2 weeks prior to the first dose of study drug(s).
3. Prior systemic therapy (e.g., chemotherapy, immunomodulatory therapy, monoclonal antibody therapy, or investigational therapy) within 4 weeks, or 5 half-lives of the drug, whichever is longer, prior to the first dose of the study drug(s).
4. History of previous treatment with EZH2 inhibition.
5. Participants currently receiving any medications or substances that are moderate or strong inducers or moderate or strong inhibitors of cytochrome P450 (CYP3A).
6. Participants currently receiving any medications or substances that are P-gp inhibitors (e.g., amiodarone, clarithromycin, diltiazem, erythromycin, ketoconazole, itraconazole, propafenone, quinidine, and verapamil).
7. Consumption of foods and beverages that are strong CYP3A inhibitors or inducers (star fruit, Seville orange, Seville orange-containing foods and beverages, grapefruit, grapefruit-containing food or beverages) within 3 days prior to the first dose of study drug(s).
8. Active immunosuppressive treatment equivalent to>10 mg of prednisone daily. Note: Short-course systemic corticosteroids (e.g., prevention/treatment for transfusion reaction) or use for a non-cancer indication (e.g., adrenal replacement) is acceptable.
9. Cardiovascular diseases with the following criteria:

   9.1 Evidence of prolongation of QT/corrected (QTc) interval (e.g., repeated episodes of QT corrected for heart rate using Fridericia s method [QTcF] >470 ms regardless of sex) (average of triplicate determinations) at screening

   9.2 Diagnosed or suspected long QT syndrome, or known family history of long QT syndrome

   9.3 History of clinically relevant ventricular arrhythmias, such as ventricular tachycardia, ventricular fibrillation, or Torsade de pointes

   9.4 Uncontrolled arrhythmia (participants with asymptomatic, controllable atrial fibrillation may be enrolled), or asymptomatic persistent ventricular tachycardia at screening

   9.5 Participant has clinically relevant bradycardia of less than 50 bpm at screening unless the participant has a pacemaker

   9.6 History of second- or third-degree heart block. Candidates with a history of heart block may be eligible if they currently have pacemakers, and have no history of fainting or clinically relevant arrhythmia with pacemakers, within 6 months prior to treatment initiation

   9.7 Myocardial infarction within 6 months prior to treatment initiation

   9.8 Angioplasty or stent graft implantation within 6 months prior to treatment initiation

   9.9 Uncontrolled angina pectoris within 6 months prior to treatment initiation

   9.10 History of New York Heart Association (NYHA), https://www.merckmanuals.com/professional/multimedia/table/new-york-heart- association-nyha-classification-of-heart-failure) Class 3 or 4 congestive heart failure

   9.11 Coronary/peripheral artery bypass graft within 6 months prior to treatment initiation

   9.12 Uncontrolled hypertension (resting systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg) at screening

   9.13 Complete left bundle branch block at screening
10. History of autoimmune disease with the exception of controlled thyroid disease, psoriasis not requiring medications, vitiligo, and alopecia.
11. Prior malignancy active within the previous 2 years except for locally curable cancer that is currently considered as cured and does not require additional Standard of Care treatment, such as cutaneous basal or squamous cell carcinoma, superficial bladder cancer, or cervical carcinoma in situ, or an incidental histological finding of prostate cancer.
12. Ongoing uncontrolled systemic bacterial, fungal, or viral infection currently requiring treatment with intravenous antibiotics, antivirals, or antifungals.
13. Pregnancy (confirmed with beta-human chorionic gonadotropin (beta-HCG) serum or urine pregnancy test performed in females of childbearing potential at screening).
14. Uncontrolled intercurrent illness or situations that would limit compliance with study requirements.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-07-09 (Actual); Primary Completion 2025-07-09 (Actual); Study Completion 2025-07-09 (Actual)

PRIMARY OUTCOMES:
Phase II: Disease control rate (DCR) | Study start until progression or 2 years after treatment initiation
  Best confirmed response in participants with PD-L1 positive (CPS >=1), HPV-negative relapsing/metatstic HNSCC treated with valemetostat and pembrolizumab compared to historical controls with pembrolizumab alone, by CT scan and brain MRI (PR+CR+SD)
Phase Ib: Safety of valemetostat in combination with pembrolizumab | Study start-30 days after last dose of study agents
  Any toxicities that occur during timeframe.
Phase Ib: Recommended phase II dose (RP2D) of valemetostat in combination with pembrolizumab | 42 days
  Number of dose limiting toxicities (DLTs) that occur within the DLT period will determine RP2D.

SECONDARY OUTCOMES:
Pharmacokinetics of valemetostat in combination with pembrolizumab | Phase Ib: C1D1, C1D8, C1D15, and C2D1Phase II: C0D1, C1D1, C1D8, C1D15, and C2D1
  Valemetostat level in blood samples collected for PK analysis
Overall survival (OS) in participants treated with valemetostat and pembrolizumab compared to historical controls with pembrolizumab alone | Study start until progression or 2 years after treatment initiation.
  Participants will be assessed for survival while on study therapy and every 9 weeks before progression / every 6 weeks after progression.
6-month progression free survival (PFS) rate in participants treated with valemetostat and pembrolizumab compared to historical controls treated with pembrolizumab alone | Phase Ib: Study start until progression or 6 months after treatment initiationPhase II: Study start until progression or 6 months after tx initiation
  Participants will be assessed for survival at 6 months after start of study, or until progression.
Progression free survival (PFS) in participants treated with valemetostat and pembrolizumab compared to historical controls with pembrolizumab alone | Phase Ib: Study start until progression or 2 years after treatment initiationPhase II: Study start until progression or 2 years after treatment initiation
  Participants will be assessed for survival until progression or 2 years after treatment start.
Clinical benefit rate (CBR) in participants treated with valemetostat and pembrolizumab compared to historical controls with pembrolizumab alone | Phase 1b: Study start until progression or 2 years after treatment initiation.Phase II: Study start until progression or 2 years after treatment initiation.
  Stable disease >= 6 months + complete response + partial response
Objective response rate (ORR) in participants treated with valemetostat and pembrolizumab compared to historical controls with pembrolizumab alone | Phase 1b: Treatment start until progression or 2 years after treatment initiation.Phase II: Treatment start until progression or 2 years after treatment initiation.
  ORR will be evaluated with periodic CT imaging.
Safety of the valemetostat and pembrolizumab combination (Phase II) | Treatment start until 30 days after last dose of study agents.
  Any toxicities identified during evaluation timeframe.

CONTACTS AND LOCATIONS:
Overall Officials: Vassiliki Saloura, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP. All collected IPD will be shared with collaborators under the terms of collaborative agreements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_001545-C.html